CLINICAL TRIAL: NCT04928287
Title: "A Randomized, Double-Blind, Single Center, Phase 2, Efficacy and Safety Study of Autologous HB-adMSCs vs Placebo for the Treatment of Patients With Parkinson's Disease"
Brief Title: Randomized, Double-Blind Clinical Trial for Parkinson's Disease (Early and Moderate)
Acronym: PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hope Biosciences Research Foundation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HBPD03
Record Dates: First submitted 2021-05-26; First posted 2021-06-16 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: A parallel study is a type of clinical study where two groups of treatments, A (HB-adMSCs) and B (Placebo), are given so that one group receives only A while another group receives only B.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study subjects, investigators and study staff will be blinded to the assigned treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HB-adMSCs (Active Comparator): Autologous Hope Biosciences adipose derived mesenchymal stem cells.
  Interventions: Biological: HB-adMSCs; Other: Placebo
- Placebo (Placebo Comparator): Sterile Saline Solution 0.9%
  Interventions: Biological: HB-adMSCs; Other: Placebo

INTERVENTIONS:
Biological: HB-adMSCs — HB-adMSCs will be administered intravenously to study participants who qualify.
  Other Names: Autologous Hope Biosciences adipose derived mesenchymal stem cells.
Other: Placebo — Placebo will be administered intravenously to study participants who qualify.
  Other Names: Sterile Saline Solution 0.9%

SUMMARY:
This is a randomized, double-blind, single center, phase 2 study to assess efficacy and safety of multiple HB-adMSCs vs Placebo for the treatment of Parkinson's disease.

The trial includes a screening period of up to 4 weeks, a 32-week treatment period, and a safety Follow-up period of 20 weeks after the last investigational product administration.

This clinical trial will be open to enroll 24 eligible participants diagnosed with Parkinson's disease. Patients' recruitment will be conducted by the study team, if eligible participants are identified based on eligibility criteria, a screening visit will be scheduled. Informed consent form will be given to the study participants and signed before any study procedures. Informed consent form will include information about the clinical trial and some aspects should be considered during this process.

ELIGIBILITY:
Inclusion Criteria:

* A study participant will be eligible for inclusion in this study only if all of the following criteria apply:

  1. Male and female participants 18 - 75 years of age.
  2. Study participant must have been diagnosed with early and/or moderate Parkinson's disease at least 6 months before study participation.
  3. Study participants must have previously banked their mesenchymal stem cells with Hope Biosciences.
  4. Study participants should be able to read, understand and to provide written consent.
  5. Voluntarily signed informed consent obtained before any clinical-trial related procedures are performed.
  6. Female study participants should not be pregnant or plan to become pregnant during study participation and for 6 months after last investigational product administration.
  7. Male participants if their sexual partners can become pregnant should use a method of contraception during study participation and for 6 months after the last administration of the investigated product.
  8. Study participant is able and willing to comply with the requirements of this clinical trial.

Exclusion Criteria:

* A study participant will not be eligible for inclusion in this clinical trial if any of the following criteria apply:

  1. Pregnancy, lactation. Women of childbearing age who are not pregnant but do not take effective contraceptive measures.
  2. Study participants with advanced Parkinson's disease described as, severe disability, wheelchair bound or bedridden.
  3. Study participant has any active malignancy, including evidence of cutaneous basal, squamous cell carcinoma or melanoma.
  4. Study participant has known alcoholic addiction or dependency or has current substance use or abuse.
  5. Study participant has 1 or more significant concurrent medical conditions (verified by medical records), including the following:

     * Poorly controlled diabetes mellitus (PCDM) defined as history of deficient standard of care treatment and/or pre-prandial glucose >130mg/dl during screening visit or post-prandial glucose >200mg/dl.
     * Medical History of Chronic kidney disease (CKD) diagnosis and/or screening results of eGFR < 59mL/min/1.73m2.
     * Presence of New York Heart Association (NYHA) Class III/IV heart failure during screening visit.
     * Any medical history of myocardial infarction in any of the different types, such as ST-elevation myocardial infarction (STEMI) or non-ST-elevated myocardial infarction (NSTEMI), coronary spasm, or unstable angina.
     * Medical history of uncontrolled high blood pressure defined as a deficient standard of care treatment and/or blood pressure > 180/120 mm/Hg during screening visit.
     * Medical history of inherited thrombophilias, recent major general surgery, (within 12 months before the Screening), lower extremity paralysis due to spinal cord injury, fracture of the pelvis, hips or femur, cancer of the lung, brain, lymphatic, gynecologic system (ovary or uterus), or gastrointestinal tract (like pancreas or stomach).
     * History of brain surgery for Parkinson's disease.
  6. Study participant has received any stem cell treatment within 6 months before first dose of investigational product other than stem cells produced by Hope Biosciences.
  7. Receiving any investigational therapy or any approved therapy for investigational use within 1 year prior first dose of the investigational product other than COVID-19 vaccines.
  8. Study participant has a laboratory abnormality during screening, including the following:

     * White blood cell count < 3000/mm3
     * Platelet count < 80,000mm3
     * Absolute neutrophil count < 1500/mm3
     * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 10 upper limit of normal (ULN) x 1.5
  9. Study participant has any other laboratory abnormality or medical condition which, in the opinion of the investigator, poses a safety risk or will prevent the subject from completing the study.
  10. Study participant is unlikely to complete the study or adhere to the study procedures.
  11. Study participant with known concurrent acute or chronic viral hepatitis B or C or human immunodeficiency virus (HIV) infection.
  12. Study participant has a previously diagnosed psychiatric condition which in the opinion of the investigator may affect self-assessments.
  13. Study participant with any systemic infection requiring treatment with antibiotics, antivirals, or antifungals within 30 days prior to first dose of the investigational product.
  14. Male study participants who plan to donate sperm during the study or within 6 months after the last dose. Female patients who plan to donate eggs or undergo in vitro fertilization treatment during the study or within 6 months after the last dose.
  15. Study participants who are determined by the Investigator to be unsuitable for study enrollment for other reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Djamchid Lotfi, MD, Principal Investigator — Hope Biosciences Stem Cell Research Foundation
Locations (1):
- Hope Biosciences Stem Cell Research Foundation, Sugar Land, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HB-adMSCs | Placebo
Started | 15 | 9
Completed | 15 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HB-adMSCs | Placebo | Total
Number analyzed (Participants) | 15 | 9 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (11.29) | 61.1 (8.99) | 60.6 (10.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 13 | 8 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 8 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 9 | 24
Height [Mean (Standard Deviation); unit: centimeter] | 174.41 (8.572) | 173.57 (10.239) | 174.09 (9.020)
Weight [Mean (Standard Deviation); unit: kilograms] | 79.56 (23.389) | 78.94 (21.280) | 79.33 (22.149)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MDS-UPDRS Part II.
Description: The MDS-UPDRS scale refers to Movement Disorder Society - Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. The MDS-UPDRS scale consists of the following 4 segments. Part II tests "Motor Aspects of Experiences of Daily Living". Each answer to the scale is evaluated by the principal investigator during the study visit. Some sections of the MDS-UPDRS scale require multiple grades assigned to each extremity.
  There are 13 items included in Part II. Part II score ranges from 0 - 52; 12 and below is mild, 30 and above is severe. Each item has 0-4 ratings: 0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe). The total score ranges from 0 to 260, with 0 indicating no disability and 260 indicating total disability. Higher values represent a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (52 points total)
Groups:
- HB-adMSCs; Placebo: Six IV infusions of autologous adipose-derived mesenchymal stem cells. Baseline laboratory values will be collected prior to first infusion and compared at following visits. Safety labs will be assessed at visit 2, 6, and 9. MDS-Unified Parkinson's Disease Rating Scale questionnaires will be assessed at all visits (Visit 1 - 9).
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (52 points total)
  Baseline | 10.00 (6.99) | 7.33 (5.15)
  Week 4 | -1.87 (2.83) | 0.11 (2.71)
  Week 8 | -2.07 (3.67) | -1.56 (3.61)
  Week 16 | -2.00 (3.23) | -0.67 (3.24)
  Week 24 | -1.33 (3.79) | -1.44 (3.00)
  Week 32 | -0.73 (3.84) | -0.44 (2.96)
  Week 42 | -0.33 (4.19) | 0.56 (2.46)
  Week 52 | 1.20 (6.61) | 1.11 (4.37)

2. Primary Outcome: Laboratory Values. CBC (% of WBC)
Description: Changes from baseline in CBC laboratory values with unit of % of white blood cell count.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: % of white blood cell count
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
% of white blood cell count
  Basophils (%) Baseline Value | 0.73 (0.947) | 0.87 (0.752)
  Basophils (%) Week 24 | 0.05 (1.196) | 0.27 (0.994)
  Basophils (%) Week 52 | 0.29 (1.92) | 0.16 (1.078)
  Eosinophils (%) Baseline Value | 1.49 (1.838) | 2.50 (1.752)
  Eosinophils (%) Week 24 | 0.24 (1.962) | 0.03 (2.492)
  Eosinophils (%) Week 52 | -0.03 (1.649) | -0.18 (2.080)
  Lymphocytes (%) Baseline Value | 32.35 (7.020) | 33.33 (9.462)
  Lymphocytes (%) Week 24 | 0.13 (9.277) | -0.51 (5.113)
  Lymphocytes (%) Week 52 | -0.06 (6.194) | -1.17 (6.361)
  Monocytes (%) Baseline value | 7.33 (2.609) | 6.72 (4.615)
  Monocytes (%) Week 24 | -0.87 (3.229) | 0.56 (4.073)
  Monocytes (%) Week 52 | -0.49 (3.670) | 1.81 (3.538)
  Neutrophils (%) Baseline Value | 56.31 (8.385) | 56.24 (8.213)
  Neutrophils (%) Week 24 | 0.43 (8.622) | -0.34 (8.259)
  Neutrophils (%) Week 52 | 0.29 (7.828) | -0.62 (4.788)

3. Primary Outcome: Laboratory Values. CBC (10^9 Cells/L)
Description: Changes from baseline in CBC laboratory values with units of 10^9 cells/L (Leukocytes, Platelets)
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
10^9 cells/L
  Platelets (10^9 cells/L) Baseline Value | 243.3 (52.38) | 209.4 (44.46)
  Platelets (10^9 cells/L) Week 24 | 9.1 (32.96) | -12.1 (12.94)
  Platelets (10^9 cells/L) Week 52 | 8.1 (23.48) | 0.8 (7.24)
  Leukocytes (10^9 cells/L) Baseline Value | 5.83 (1.891) | 5.47 (1.267)
  Leukocytes (10^9 cells/L) Week 24 | -0.36 (1.640) | -0.08 (1.335)
  Leukocytes (10^9 cells/L) Week 52 | 0.09 (1.615) | -0.11 (0.885)

4. Primary Outcome: Laboratory Values. CBC (10^12 Cells/L)
Description: Changes from baseline in CBC laboratory values with units of 10^12 cells/L.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
10^12 cells/L
  Erythrocytes (10^12 cells /L) Baseline Value | 4.425 (0.5909) | 4.723 (0.4661)
  Erythrocytes (10^12 cells/L ) Week 24 | 0.021 (0.2671) | 0.129 (0.2073)
  Erythrocytes (10^12 cells/L ) Week 52 | 0.109 (0.3503) | 0.024 (0.1843)

5. Primary Outcome: Laboratory Values. CBC (pg)
Description: Changes from baseline in CBC laboratory values with unit of pg.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
pg
  Ery. Mean Corpuscular Hemoglobin Baseline Value | 30.80 (1.838) | 30.08 (1.949)
  Ery. Mean Corpuscular Hemoglobin Week 24 | 0.01 (0.816) | -0.12 (0.616)
  Ery. Mean Corpuscular Hemoglobin Week 52 | -0.06 (1.005) | -0.32 (0.874)

6. Primary Outcome: Laboratory Values. CBC (fL)
Description: Changes from baseline in CBC laboratory values with unit of fL.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
fL
  Ery. Mean Corpuscular Volume (fL) Baseline value | 90.83 (4.404) | 88.30 (3.508)
  Ery. Mean Corpuscular Volume (fL) Week 24 | -0.85 (1.968) | -0.46 (1.074)
  Ery. Mean Corpuscular Volume (fL) Week 52 | 0.12 (2.034) | 0.53 (1.111)

7. Primary Outcome: Laboratory Values. CBC (g/dL)
Description: Changes from baseline in CBC laboratory values with unit of g/dL.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
g/dL
  Ery. Mean Corpuscular HGB Concentration (g/dL) Baseline Value | 33.89 (0.718) | 34.03 (0.930)
  Ery. Mean Corpuscular HGB Concentration (g/dL) Week 24 | 0.34 (0.741) | 0.06 (0.781)
  Ery. Mean Corpuscular HGB Concentration (g/dL) Week 52 | -0.07 (1.306) | -0.54 (1.242)
  Hemoglobin (g/dL) Baseline Value | 13.57 (1.435) | 14.16 (1.041)
  Hemoglobin (g/dL) Week 24 | 0.09 (0.798) | 0.33 (0.561)
  Hemoglobin (g/dL) Week 52 | 0.33 (0.893) | -0.06 (0.652)

8. Primary Outcome: Laboratory Values. CBC (% Difference in Volume and Size of RBC)
Description: Changes from baseline in CBC laboratory values with unit of % difference in volume and size of RBC
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: % difference in volume and size of RBC
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
% difference in volume and size of RBC
  Erythrocytes Distribution Width (%) Baseline Value | 12.39 (0.491) | 12.64 (0.590)
  Erythrocytes Distribution Width (%) Week 24 | 0.33 (0.339) | 0.68 (1.394)
  Erythrocytes Distribution Width (%) Week 52 | 0.16 (0.364) | 0.22 (0.233)

9. Primary Outcome: Laboratory Values. CBC (% of Total Blood Cell Count)
Description: Changes from baseline in CBC laboratory values with unit of % of total blood cell count.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: % of total blood cell count
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
% of total blood cell count
  Hematocrit (%) Baseline Value | 40.01 (4.348) | 41.63 (3.403)
  Hematocrit (%) Week 24 | -0.15 (2.143) | 0.91 (1.900)
  Hematocrit (%) Week 52 | 1.13 (3.297) | 0.44 (1.519)

10. Primary Outcome: Vital Signs. - Blood Pressure (mmHg)
Description: Change from baseline in Blood Pressure.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
mmHg
  Systolic Baseline Value | 129.0 (14.63) | 135.6 (9.53)
  Systolic Week 4 | -1.9 (11.78) | -8.7 (6.22)
  Systolic Week 8 | -5.9 (10.82) | -6.3 (7.12)
  Systolic Week 16 | -3.9 (15.76) | -9.2 (5.93)
  Systolic Week 24 | -5.1 (17.33) | -6.0 (11.90)
  Systolic Week 32 | -5.8 (12.01) | -8.0 (11.11)
  Systolic Week 42 | -4.3 (18.52) | -11.6 (11.70)
  Systolic Week 52 | -5.9 (14.19) | -7.0 (11.27)
  Diastolic Baseline Value | 79.7 (10.73) | 79.8 (5.74)
  Diastolic Week 4 | -1.3 (8.38) | -2.3 (5.34)
  Diastolic Week 8 | -2.5 (7.59) | -1.0 (6.84)
  Diastolic Week 16 | -2.3 (9.42) | -3.8 (6.67)
  Diastolic Week 24 | -3.1 (8.56) | -3.6 (8.31)
  Diastolic Week 32 | -1.9 (7.80) | -1.1 (6.05)
  Diastolic Week 42 | -1.2 (11.48) | -4.0 (6.30)
  Diastolic Week 52 | 0.3 (8.09) | -0.7 (7.05)

11. Primary Outcome: Weight in kg.
Description: Change from baseline in Weight in kg.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
kg
  Baseline Value | 79.65 (23.298) | 78.94 (21.280)
  Week 4 | 0.43 (1.551) | 0.33 (1.038)
  Week 8 | 1.75 (8.868) | 0.44 (0.981)
  Week 16 | 1.73 (9.009) | 1.39 (2.354)
  Week 24 | -1.12 (2.995) | 1.04 (2.222)
  Week 32 | -0.97 (3.580) | 1.02 (2.790)
  Week 42 | -2.11 (5.441) | 3.48 (7.931)
  Week 52 | -1.77 (5.046) | 0.60 (2.926)

12. Primary Outcome: Laboratory Values. CMP (mg/dL)
Description: Change from baseline in CMP values with units of mg/dL
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
mg/dL
  Bilirubin (mg/dL) Baseline Value | 0.46 (0.150) | 0.46 (0.124)
  Bilirubin (mg/dL) Week 24 | 0.03 (0.139) | 0.10 (0.212)
  Bilirubin (mg/dL) Week 52 | 0.05 (0.177) | 0.09 (0.262)
  Calcium (mg/dL) Baseline Value | 9.63 (0.410) | 9.56 (0.357)
  Calcium (mg/dL) Week 24 | -0.06 (0.374) | 0.12 (0.387)
  Calcium (mg/dL) Week 52 | 0.09 (0.252) | -0.07 (0.442)
  Creatinine (mg/dL) Baseline Value | 0.898 (0.1243) | 0.910 (0.2579)
  Creatinine (mg/dL) Week 24 | -0.016 (0.0755) | -0.019 (0.2204)
  Creatinine (mg/dL) Week 52 | -0.031 (0.1058) | -0.082 (0.1664)
  Glucose (mg/dL) Baseline Value | 99.7 (20.78) | 100.4 (16.96)
  Glucose (mg/dL) Week 24 | 3.7 (25.95) | 10.0 (24.17)
  Glucose (mg/dL) Week 52 | 0.1 (24.14) | 0.4 (20.88)
  Urea Nitrogen (mg/dL) Baseline valuse | 16.5 (3.83) | 15.4 (4.10)
  Urea Nitrogen (mg/dL) Week 24 | 0.4 (2.61) | 1.4 (3.05)
  Urea Nitrogen (mg/dL) Week 52 | 0.0 (3.44) | 1.7 (3.84)

13. Primary Outcome: Laboratory Values. CMP (g/dL)
Description: Changes from baseline in CMP laboratory values with units of g/dL
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
g/dL
  Albumin (g/dL) Baseline Value | 4.51 (0.225) | 4.53 (0.278)
  Albumin (g/dL) Week 24 | -0.03 (0.246) | 0.08 (0.222)
  Albumin (g/dL) Week 52 | -0.01 (0.267) | -0.04 (0.167)
  Globulin (g/dL) Baseline Value | 2.61 (0.328) | 2.42 (0.497)
  Globulin (g/dL) Week 24 | -0.04 (0.206) | 0.07 (0.173)
  Globulin (g/dL) Week 52 | -0.01 (0.264) | -0.09 (0.176)
  Protein (g/dL) Baseline Value | 7.11 (0.391) | 6.96 (0.520)
  Protein (g/dL) Week 24 | -0.07 (0.406) | 0.14 (0.300)
  Protein (g/dL) Week 52 | -0.03 (0.394) | -0.13 (0.250)

14. Primary Outcome: Laboratory Values. CMP (IU/L)
Description: Changes from baseline in CMP laboratory values with units of IU/L.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
IU/L
  Alkaline Phosphatase (IU/L) Baseline Value | 63.9 (17.33) | 75.7 (17.79)
  Alkaline Phosphatase (IU/L) Week 24 | 2.3 (10.25) | 3.7 (11.81)
  Alkaline Phosphatase (IU/L) Week 52 | 2.3 (12.97) | -0.1 (6.41)
  Alanine Aminotransferase (IU/L) Baseline Value | 14.13 (8.007) | 18.31 (11.221)
  Alanine Aminotransferase (IU/L) Week 24 | -0.13 (6.611) | -2.43 (8.754)
  Alanine Aminotransferase (IU/L) Week 52 | 1.13 (5.657) | 0.68 (8.277)
  Aspartate Aminotransferase (IU/L) Baseline Value | 20.3 (6.80) | 20.3 (6.32)
  Aspartate Aminotransferase (IU/L) Week 24 | 0.0 (4.34) | -0.1 (3.10)
  Aspartate Aminotransferase (IU/L) Week 52 | 3.3 (9.52) | 0.8 (3.77)

15. Primary Outcome: Laboratory Values. CMP (mL/Min/1.73m^2)
Description: Changes from baseline in CMP laboratory values with units of mL/min/1.73m^2.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
mL/min/1.73m^2
  Glomerular Filtration Rate (mL/min/1.73m^2) Baseline Value | 80.7 (11.26) | 81.9 (16.07)
  Glomerular Filtration Rate (mL/min/1.73m^2) Week 24 | 4.6 (6.57) | 5.7 (19.04)
  Glomerular Filtration Rate (mL/min/1.73m^2) Week 52 | 6.4 (9.19) | 9.9 (14.50)

16. Primary Outcome: Laboratory Values. CMP (mmol/L)
Description: Changes from baseline in CMP laboratory values with units of mmol/L.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
mmol/L
  Chloride (mmol/L) Baseline Value | 104.5 (1.41) | 104.4 (2.19)
  Chloride (mmol/L) Week 24 | 0.5 (1.73) | -2.0 (1.80)
  Chloride (mmol/L) Week 52 | -0.3 (2.31) | -0.1 (2.42)
  Carbon Dioxide (mmol/L) Baseline Value | 25.7 (2.28) | 26.2 (2.54)
  Carbon Dioxide (mmol/L) Week 24 | -0.9 (2.13) | -1.2 (2.39)
  Carbon Dioxide (mmol/L) Week 52 | 0.0 (1.89) | -0.2 (2.22)
  Potassium (mmol/L) Baseline Value | 4.29 (0.287) | 4.31 (0.190)
  Potassium (mmol/L) Week 24 | 0.04 (0.333) | -0.01 (0.220)
  Potassium (mmol/L) Week 52 | 0.02 (0.273) | -0.01 (0.209)
  Sodium (mmol/L) Baseline Value | 141.5 (1.88) | 142.2 (1.64)
  Sodium (mmol/L) Week 24 | -0.1 (1.98) | -1.9 (1.54)
  Sodium (mmol/L) Week 52 | 0.1 (2.37) | -1.0 (2.00)

17. Primary Outcome: Laboratory Values. CMP (Ratio: Albumin (g/dL) to Calc. Globulin (g/dL))
Description: Changes from baseline in CMP laboratory values with units of Ratio: Albumin(g/dL) to Calc. Globulin(g/dL)
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: Ratio: Albumin(g/dL) to Globulin(g/dL)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
Ratio: Albumin(g/dL) to Globulin(g/dL)
  Albumin/Globulin (RATIO) Baseline Value | 1.75 (0.236) | 1.96 (0.467)
  Albumin/Globulin (RATIO) Week 24 | 0.03 (0.118) | -0.03 (0.150)
  Albumin/Globulin (RATIO) Week 52 | 0.02 (0.214) | 0.03 (0.166)

18. Primary Outcome: Laboratory Values. CMP (Ratio: Urea Nitrogen (mg/dL) to Creatinine (mg/dL))
Description: Changes from baseline in CMP laboratory values with units of Ratio: Urea Nitrogen (mg/dL) to Creatinine (mg/dL)
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: Ratio:Urea nit.(mg/dL) /creatinin(mg/dL)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
Ratio:Urea nit.(mg/dL) /creatinin(mg/dL)
  Urea Nitrogen/Creatinine (RATIO) Baseline Value | 18.5 (4.49) | 18.0 (5.07)
  Urea Nitrogen/Creatinine (RATIO) Week 24 | 1.1 (3.27) | 1.1 (5.73)
  Urea Nitrogen/Creatinine (RATIO) Week 52 | 0.8 (3.91) | 4.4 (9.00)

19. Primary Outcome: Laboratory Values. Coagulation Panel (Seconds)
Description: Changes from baseline in Coagulation Panel values with units of seconds.
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
seconds
  Prothrombin Time (sec) Baseline Value | 13.20 (0.332) | 13.22 (0.814)
  Prothrombin Time (sec) Week 24 | 0.07 (0.505) | -0.08 (0.604)
  Prothrombin Time (sec) Week 52 | 0.13 (0.294) | -0.08 (0.751)
  Partial Thromboplastin Time (sec) Baseline Value | 29.47 (2.446) | 31.00 (7.112)
  Partial Thromboplastin Time (sec) Week 24 | 0.42 (1.026) | -1.47 (5.437)
  Partial Thromboplastin Time (sec) Week 52 | 0.11 (1.235) | -1.37 (6.275)

20. Primary Outcome: Laboratory Values. Coagulation Panel (Ratio: Prothrombin Time (Seconds) / Mean Normal Prothrombin Time (Seconds))
Description: Changes from baseline in Coagulation laboratory values with units of Ratio: Prothrombin time (seconds) / Mean normal prothrombin time (seconds).
Time Frame: Baseline (Week 0), Week 24, and End of Study (Week 52)
Measure: Mean (Standard Deviation); unit: Ratio: PT (seconds) / MNPT (seconds)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
Ratio: PT (seconds) / MNPT (seconds)
  Prothrombin Intl. Normalized Ratio (RATIO) Baseline Value | 0.97 (0.049) | 0.96 (0.073)
  Prothrombin Intl. Normalized Ratio (RATIO) Week 24 | 0.01 (0.074) | 0.02 (0.067)
  Prothrombin Intl. Normalized Ratio (RATIO) Week 52 | 0.01 (0.035) | -0.00 (0.050)

21. Primary Outcome: Vital Signs. - Respiratory Rate (Breaths Per Minute)
Description: Changes from Baseline in Respiratory Rate.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
breaths/minute
  Baseline Value | 16.3 (0.70) | 16.0 (0.00)
  Week 4 | 0 (0) | 0.2 (0.67)
  Week 8 | 0.1 (1.19) | 0.2 (0.67)
  Week 16 | -0.1 (0.52) | 0.0 (0.0)
  Week 24 | 0.1 (0.92) | 0.4 (0.88)
  Week 32 | 0.7 (0.98) | 0.7 (1.00)
  Week 42 | 0.4 (1.12) | 0.4 (0.88)
  Week 52 | 0.3 (0.70) | 0.7 (1.00)

22. Primary Outcome: Vital Signs. - Heart Rate (Beats Per Minute)
Description: Change from baseline in Heart Rate.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
beats/minute
  Baseline Value | 70.7 (10.80) | 69.8 (9.61)
  Week 4 | -1.3 (6.27) | 1.9 (8.72)
  Week 8 | -2.1 (6.46) | 0.4 (4.36)
  Week 16 | -2.1 (8.46) | 3.4 (13.18)
  Week 24 | 4.3 (9.30) | 1.1 (6.95)
  Week 32 | 3.8 (6.61) | 1.7 (3.77)
  Week 42 | 3.5 (6.22) | -0.3 (7.68)
  Week 52 | 5.3 (10.54) | 0.7 (4.21)

23. Primary Outcome: Vital Signs. - Body Temperature (Celsius )
Description: Change from baseline in Body Temperature.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
Celsius
  Baseline Value | 36.59 (0.245) | 36.54 (0.133)
  Week 4 | 0.09 (0.351) | -0.03 (0.194)
  Week 8 | -0.02 (0.288) | -0.11 (0.232)
  Week 16 | 0.09 (0.275) | -0.01 (0.247)
  Week 24 | 0.05 (0.409) | -0.07 (0.316)
  Week 32 | 0.12 (0.334) | 0.11 (0.330)
  Week 42 | 0.13 (0.324) | -0.06 (0.350)
  Week 52 | 0.05 (0.342) | 0.03 (0.296)

24. Secondary Outcome: Change From Baseline in MDS-UPDRS Part I.
Description: The MDS-UPDRS scale refers to Movement Disorder Society - Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. Part I tests "Nonmotor experiences of daily living". Non-Motor Aspects of Experiences of Daily Living (nM-EDL), including complex behaviors such as, cognitive impairment, hallucinations and psychosis, depressed mood, anxious mood, apathy, features of dopamine dysregulation syndrome, sleep problems, daytime sleepiness, pain and other sensations, urinary problems, constipation problems, light headedness on standing and fatigue.
  There are 13 items included in Part I. Part I score ranges from 0 - 52; 10 and below is mild, 22 and above is severe. Each item has 0-4 ratings:0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe). The total score ranges from 0 to 260, with 0 indicating no disability and 260 indicating total disability. Higher values represent a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (52 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (52 points total)
  Baseline Value | 8.73 (5.95) | 6.78 (4.94)
  Week 4 | -1.47 (2.50) | 0.33 (2.83)
  Week 8 | -1.67 (3.02) | -0.33 (2.96)
  Week 16 | -2.53 (3.80) | 0.33 (2.92)
  Week 24 | -1.40 (3.94) | 0.22 (3.11)
  Week 32 | -2.07 (4.11) | -0.33 (3.67)
  Week 42 | -0.87 (4.26) | 1.56 (3.75)
  Week 52 | -0.47 (4.27) | 0.78 (4.15)

25. Secondary Outcome: Change From Baseline in MDS-UPDRS Part III.
Description: The MDS-UPDRS scale refers to Movement Disorder Society - Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. Part III tests "Motor examination". Motor Examination includes speech, facial expression, rigidity, finger and hand movement, pronation-supination movements of hands, toe tapping, leg agility, arising from chair, gait, freezing of gait, postural stability, posture, global spontaneity of movement, postural tremor of the hands, kinetic tremor of the hands, rest tremor amplitude, constancy of rest tremor, dyskinesias impact and Hoehn and Yahr stage.
  There are 18 items included in Part III. Part III score ranges from 0 - 132; 32 and below is mild, 59 and above is severe. Each item has 0-4 ratings:0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe). The total score ranges from 0 to 260, with 0 indicating no disability and 260 indicating total disability. Higher values represent a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (132 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (132 points total)
  Baseline Value | 26.27 (12.76) | 20.56 (8.35)
  Week 4 | -5.33 (8.72) | -0.33 (10.74)
  Week 8 | -8.33 (12.73) | -1.78 (9.85)
  Week 16 | -8.13 (13.52) | -0.22 (11.63)
  Week 24 | -10.07 (16.50) | -2.78 (12.25)
  Week 32 | -11.27 (13.82) | -4.33 (8.93)
  Week 42 | -8.47 (15.25) | -3.56 (11.28)
  Week 52 | -9.07 (14.23) | -4.11 (6.31)

26. Secondary Outcome: Change From Baseline in MDS-UPDRS Part IV.
Description: The MDS-UPDRS scale refers to Movement Disorder Society - Unified Parkinson Disease Rating Scale, and it is a rating tool used to gauge the course of Parkinson's disease in patients. Part IV tests "Motor Complications", including time spent with dyskinesias and others.
  There are 6 items included in Part IV. Part IV score ranges from 0 - 24; 4 and below is mild, 13 and above is severe. Each item has 0-4 ratings:0 (normal), 1 (slight), 2 (mild), 3 (moderate), and 4 (severe). The total score ranges from 0 to 260, with 0 indicating no disability and 260 indicating total disability. Higher values represent a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (24 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (24 points total)
  Baseline Value | 2.67 (3.77) | 3.56 (2.30)
  Week 4 | -0.67 (2.19) | -0.33 (1.94)
  Week 8 | -0.87 (1.51) | -0.44 (2.46)
  Week 16 | -1.00 (1.93) | -1.00 (1.94)
  Week 24 | -1.87 (2.88) | 0.00 (2.00)
  Week 32 | -2.20 (3.28) | -0.67 (2.45)
  Week 42 | -0.80 (2.01) | -1.11 (1.83)
  Week 52 | -1.07 (3.10) | -1.67 (1.66)

27. Secondary Outcome: Change From Baseline in Neuro-QOL. - Communication
Description: Communication - Short Form
  Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The communication short form has 5 questions regarding communicative abilities of the patient, and each question ranges from 0 points to 5 points (making the total 25 points). A higher score represents a better outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (25 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (25 points total)
  Baseline Value | 22.87 (2.83) | 21.78 (4.55)
  Week 4 | 0.40 (0.83) | 2.00 (4.66)
  Week 8 | 0.53 (1.92) | 1.33 (2.92)
  Week 16 | 0.67 (1.45) | 1.56 (4.69)
  Week 24 | 0.00 (0.85) | 1.89 (4.31)
  Week 32 | 0.27 (1.22) | 1.89 (4.59)
  Week 42 | 0.00 (0.76) | 1.78 (4.68)
  Week 52 | -0.60 (2.67) | 1.00 (4.61)

28. Secondary Outcome: Change From Baseline in Neuro-QOL. - Social Roles and Activities
Description: Ability to Participate in Social Roles and Activities - Short Form
  Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Ability to Participate in Social Roles and Activities" short form has 8 questions regarding social abilities of the patient (familial and friend relationships), and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a better outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 36.00 (4.68) | 35.22 (5.14)
  Week 4 | 0.93 (2.62) | 1.00 (5.15)
  Week 8 | 0.47 (3.04) | 1.22 (5.38)
  Week 16 | 1.73 (4.13) | 0.56 (6.84)
  Week 24 | -2.27 (8.03) | 2.33 (6.26)
  Week 32 | -0.40 (2.69) | 0.78 (5.12)
  Week 42 | 0.13 (4.70) | 0.56 (6.44)
  Week 52 | -1.93 (7.16) | 0.33 (7.09)

29. Secondary Outcome: Changes From Baseline in Neuro-QOL. - Anxiety
Description: Anxiety - Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Anxiety" short form has 8 questions regarding the anxiety level of the patient (inquiring about level of uneasiness and worry), and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 17.87 (6.51) | 14.11 (4.11)
  Week 4 | -1.40 (3.74) | -1.00 (2.60)
  Week 8 | -2.40 (2.35) | -1.44 (2.92)
  Week 16 | -3.07 (4.22) | -0.22 (4.38)
  Week 24 | -2.33 (5.45) | -1.67 (3.57)
  Week 32 | -1.80 (5.10) | -1.44 (4.50)
  Week 42 | -2.07 (5.68) | -2.00 (4.06)
  Week 52 | -2.00 (4.36) | -1.56 (3.84)

30. Secondary Outcome: Change From Baseline in Neuro-QOL. - Depression
Description: Depression - Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Depression" short form has 8 questions regarding the depression level of the patient, and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 12.40 (4.81) | 9.89 (2.26)
  Week 4 | -2.27 (3.39) | 0.11 (2.15)
  Week 8 | -2.00 (3.44) | -0.11 (3.26)
  Week 16 | -2.60 (3.36) | 0.44 (1.24)
  Week 24 | -1.00 (5.44) | 0.00 (1.32)
  Week 32 | -1.47 (3.91) | 1.56 (3.97)
  Week 42 | -1.80 (4.97) | 0.11 (1.96)
  Week 52 | -1.40 (4.32) | 1.11 (2.98)

31. Secondary Outcome: Change From Baseline in Neuro-QOL. - Dyscontrol
Description: Emotional and Behavioral Dyscontrol - Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Dyscontrol" short form has 8 questions regarding the emotional and behavioral dyscontrol level of the patient, and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 13.47 (5.36) | 10.89 (3.37)
  Week 4 | -0.33 (3.56) | -0.11 (2.47)
  Week 8 | -1.07 (1.87) | -0.67 (2.55)
  Week 16 | -1.67 (3.52) | 0.22 (3.70)
  Week 24 | -1.07 (2.99) | -1.11 (2.20)
  Week 32 | 0.20 (4.35) | -0.78 (2.86)
  Week 42 | -0.73 (4.01) | -0.78 (2.64)
  Week 52 | -0.93 (3.17) | -0.78 (2.59)

32. Secondary Outcome: Changes From Baseline in Neuro-QOL. - Fatigue
Description: Fatigue - Short Form Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Fatigue" short form has 8 questions regarding the Fatigue level of the patient, and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 16.67 (7.90) | 14.11 (4.46)
  Week 4 | -1.73 (3.10) | 0.11 (3.69)
  Week 8 | -1.67 (3.46) | -1.11 (4.86)
  Week 16 | -2.40 (4.75) | 1.67 (5.63)
  Week 24 | -1.13 (6.24) | 0.33 (4.82)
  Week 32 | -2.00 (4.99) | 0.11 (7.17)
  Week 42 | -0.93 (6.09) | -0.33 (5.85)
  Week 52 | 1.47 (5.04) | 0.67 (5.89)

33. Secondary Outcome: Change From Baseline in Neuro-QOL. - Mobility
Description: Lower Extremity Function (Mobility) - Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Mobility" short form has 8 questions regarding the Lower Extremity Function (Mobility) level of the patient, and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 37.00 (3.09) | 38.22 (3.11)
  Week 4 | -0.53 (1.88) | 0.33 (3.08)
  Week 8 | -0.33 (3.46) | 0.22 (2.68)
  Week 16 | 0.53 (3.50) | 1.22 (2.91)
  Week 24 | 0.13 (3.14) | 0.11 (3.98)
  Week 32 | -0.07 (2.79) | -0.33 (4.50)
  Week 42 | -0.53 (2.88) | -0.33 (3.43)
  Week 52 | -1.67 (5.00) | -0.67 (2.96)

34. Secondary Outcome: Change From Baseline in Neuro-QOL. - Well-Being
Description: Positive Affect and Well-Being - Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Positive Affect and Well-Being" short form has 8 questions regarding the well-being level of the patient, and each question ranges from 0 points to 5 points (making the total 45 points). A higher score represents a better outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (45 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (45 points total)
  Baseline Value | 36.87 (5.22) | 39.00 (4.39)
  Week 4 | 3.00 (3.23) | -1.22 (5.21)
  Week 8 | 2.73 (2.94) | 0.33 (5.05)
  Week 16 | 4.33 (5.05) | -0.44 (4.33)
  Week 24 | 0.80 (4.63) | 1.00 (5.57)
  Week 32 | 1.67 (3.89) | -1.89 (5.53)
  Week 42 | 1.67 (5.60) | 0.00 (4.50)
  Week 52 | 2.67 (4.42) | -1.78 (8.97)

35. Secondary Outcome: Change From Baseline in Neuro-QOL. - Sleep
Description: Sleep Disturbance - Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Sleep disturbance" short form has 8 questions regarding the sleep level of the patient, and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 16.20 (6.32) | 14.33 (4.74)
  Week 4 | -2.33 (4.45) | -1.89 (2.98)
  Week 8 | -1.73 (5.27) | -1.89 (3.55)
  Week 16 | -2.60 (5.74) | -0.11 (3.86)
  Week 24 | -3.27 (5.50) | -1.22 (3.87)
  Week 32 | -3.00 (5.73) | -2.33 (4.95)
  Week 42 | -1.93 (6.12) | -1.22 (5.38)
  Week 52 | -1.93 (5.04) | -1.67 (5.41)

36. Secondary Outcome: Change From Baseline in Neuro-QOL. - Fine Motor
Description: Upper Extremity Function (Fine Motor, ADL) - Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Upper Extremity Function (Fine Motor, ADL)" short form has 8 questions regarding the fine motor levels of the patient, and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a better outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 36.07 (4.37) | 37.33 (2.65)
  Week 4 | 0.80 (2.11) | 1.67 (2.50)
  Week 8 | 0.47 (1.68) | 1.11 (1.69)
  Week 16 | 1.93 (3.10) | 0.78 (2.17)
  Week 24 | 0.87 (2.33) | 1.22 (1.48)
  Week 32 | 0.40 (2.56) | 0.56 (1.42)
  Week 42 | -0.60 (4.14) | 0.44 (1.42)
  Week 52 | -0.53 (3.09) | 0.67 (1.50)

37. Secondary Outcome: Change From Baseline in Neuro-QOL. - Stigma
Description: Stigma-Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Stigma" short form has 8 questions regarding the stigma levels of the patient, and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 12.33 (4.48) | 12.00 (3.87)
  Week 4 | -1.20 (3.71) | -1.22 (2.82)
  Week 8 | -0.67 (3.75) | -1.44 (2.46)
  Week 16 | -1.27 (3.49) | -0.33 (2.92)
  Week 24 | -1.40 (3.52) | -1.22 (2.49)
  Week 32 | -0.67 (3.75) | -0.89 (1.36)
  Week 42 | -1.87 (3.89) | -0.56 (1.81)
  Week 52 | -0.93 (3.84) | -1.89 (2.47)

38. Secondary Outcome: Change From Baseline in Neuro-QOL. - Social Roles
Description: Satisfaction with Social Roles and Activities - Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Satisfaction with Social Roles and Activities" short form has 8 questions regarding the satisfaction levels of the patient, and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a better outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 30.47 (5.68) | 33.78 (5.31)
  Week 4 | 3.27 (7.39) | 1.22 (4.71)
  Week 8 | 2.87 (6.57) | 1.89 (4.99)
  Week 16 | 3.87 (8.74) | -0.44 (8.16)
  Week 24 | 2.27 (6.31) | -1.67 (7.81)
  Week 32 | 1.53 (8.42) | 1.56 (3.68)
  Week 42 | 1.53 (9.03) | 1.67 (4.66)
  Week 52 | 1.20 (6.65) | 0.44 (3.64)

39. Secondary Outcome: Change From Baseline in Neuro-QOL. - Cognition
Description: Cognition Function- Short Form Neuro-QoL (Quality of Life in Neurological Disorders) is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The "Cognition Function" short form has 8 questions regarding the cognition function levels of the patient, and each question ranges from 0 points to 5 points (making the total 40 points). A higher score represents a better outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (40 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (40 points total)
  Baseline Value | 33.47 (6.21) | 33.67 (5.68)
  Week 4 | 2.53 (3.29) | 1.44 (2.55)
  Week 8 | 1.33 (3.74) | 0.89 (2.89)
  Week 16 | 2.80 (5.05) | 1.00 (2.18)
  Week 24 | 2.87 (4.98) | 2.00 (3.04)
  Week 32 | 0.73 (7.46) | 2.44 (3.88)
  Week 42 | 0.87 (5.91) | 2.44 (4.33)
  Week 52 | 0.47 (7.12) | 1.56 (4.36)

40. Secondary Outcome: Change From Baseline in Parkinson's Disease Fatigue Scale (PFS-16).
Description: The Parkinson's disease fatigue scale (PFS-16) is an 16 question assessment that measures the level of fatigue in patients diagnosed with Parkinson's disease. Each question has 5 answer choices established as "strongly disagree", "disagree", "do not agree or disagree", "agree", and "strongly agree", which are scored as 1 to 5, respectively, making the total score from 16 to 80 points. Higher score represents a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (80 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (80 points total)
  Baseline Value | 37.20 (18.18) | 34.11 (15.21)
  Week 4 | -0.73 (10.59) | -8.33 (9.46)
  Week 8 | 0.20 (5.23) | -4.33 (12.25)
  Week 16 | -3.40 (7.70) | -2.33 (9.79)
  Week 24 | -2.33 (10.38) | -4.11 (8.45)
  Week 32 | -3.00 (12.58) | -3.56 (12.08)
  Week 42 | -1.00 (11.43) | -4.11 (8.34)
  Week 52 | 2.67 (5.29) | -2.89 (11.77)

41. Secondary Outcome: Change From Baseline in Parkinson's Disease Questionnaire (PDQ-39).
Description: The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. Items are grouped into eight scales that are scored by expressing summed item scores as a percentage score ranging between 0 and 100. The final reported score (summary index) is calculated by averaging the 8 scaled scores. Higher score represents a worse outcome.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (100 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (100 points total)
  Baseline Value | 28.13 (20.20) | 18.67 (12.18)
  Week 4 | -4.87 (10.03) | -2.78 (8.71)
  Week 8 | -4.67 (14.36) | -4.33 (12.49)
  Week 16 | -6.60 (14.25) | -0.11 (14.34)
  Week 24 | -7.07 (13.25) | 0.11 (14.38)
  Week 32 | -6.93 (12.48) | -2.67 (9.75)
  Week 42 | -4.93 (13.41) | -2.33 (12.76)
  Week 52 | -0.33 (16.60) | 0.33 (12.31)

42. Secondary Outcome: Change From Baseline in Total Visual Analog Scale
Description: Visual Analog Scale for Pain and Muscle Spasm. The pain and muscle spasm VAS is a unidimensional measure of pain/ muscle spasm intensity, used to record patients' pain progression and muscle spasm progression, or compare pain and muscle spasm severity between patients with similar conditions. Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark summed with the distance (mm) on the 10-cm line between the "no muscle spasm" anchor and the patient's mark, providing a range of scores from 0-200. A higher score indicates greater pain/spasm intensity.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: score on a scale (200 points total)
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
score on a scale (200 points total)
  Baseline Value | 35.93 (37.75) | 19.89 (21.80)
  Week 4 | -5.33 (32.87) | 2.89 (16.80)
  Week 8 | -8.27 (10.92) | -3.33 (10.69)
  Week 16 | -3.53 (20.78) | 16.11 (68.18)
  Week 24 | -11.0 (37.63) | 6.78 (29.85)
  Week 32 | -15.13 (37.05) | 9.22 (34.82)
  Week 42 | -7.80 (31.93) | 9.89 (22.65)
  Week 52 | -6.73 (21.53) | -10.00 (16.41)

43. Secondary Outcome: Change From Baseline in Dosage of Carbidopa/Levodopa
Description: Dosage of medications.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
mg
  Baseline Value | 439.3 (599.96) | 285.6 (273.92)
  Week 4 | 0 (0) | 0 (0)
  Week 8 | 0 (0) | 0 (0)
  Week 16 | 20. (77.46) | 11.1 (33.33)
  Week 24 | 0 (0) | 11.1 (33.33)
  Week 32 | 0 (0) | 11.1 (33.33)
  Week 42 | 0 (0) | 36.1 (54.65)
  Week 52 | -10.0 (89.04) | 47.2 (75.46)

44. Secondary Outcome: Change From Baseline in Vital Signs. - Oxygen Saturation.
Description: Changes in Oxygen Saturation.
Time Frame: Baseline through Week 32, Follow-up at week 42 and End of Study at week 52
Measure: Mean (Standard Deviation); unit: percent of oxygen
Arm/Group | HB-adMSCs | Placebo
Number analyzed (Participants) | 15 | 9
percent of oxygen
  Baseline Value | 97.8 (1.01) | 97.6 (1.74)
  Week 4 | -0.2 (2.14) | -1.0 (2.65)
  Week 8 | 0.2 (1.08) | 0.6 (1.42)
  Week 16 | 0.1 (0.88) | -0.2 (1.72)
  Week 24 | -0.5 (0.83) | 0.1 (1.05)
  Week 32 | -0.3 (0.82) | 0.3 (1.73)
  Week 42 | -0.6 (1.18) | 0.0 (1.41)
  Week 52 | -0.7 (1.50) | 0.3 (1.00)

ADVERSE EVENTS:
Time Frame: Week 0 (Infusion 1) through Week 52 (End of Study)
Arm/Group | HB-adMSCs | Placebo
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/9
Other Adverse Events (participants affected / at risk) | 15/15 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HB-adMSCs (N=15) | Placebo (N=9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HB-adMSCs (N=15) | Placebo (N=9)
Headache (Nervous system disorders) | 5 (11) | 1 (6)
Tremor (Nervous system disorders) | 1 (1) | 4 (6)
Balance Difficulty (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (3) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Frozen Gait (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Near Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (5) | 1 (1)
Influenza-like symptoms (General disorders) | 2 (3) | 1 (1)
Ankle edema (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Drug Ineffective (General disorders) | 0 (0) | 1 (1)
Feverish (General disorders) | 1 (2) | 0 (0)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Joint Pain (General disorders) | 1 (1) | 0 (0)
Limb Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Stiff Neck (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Swollen ankles (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hazy Vision (Eye disorders) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Eyelid twitching (Eye disorders) | 1 (1) | 0 (0)
Eyes heavy feeling of (Eye disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (3) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Increased salivation (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 virus test positive (Investigations) | 0 (0) | 1 (1)
Hypercholesterolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Kidney Stone (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Eye laser surgery (Surgical and medical procedures) | 1 | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT04928287/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT04928287/SAP_001.pdf